CLINICAL TRIAL: NCT02718664
Title: Food-effect Study on Uracil and Dihydrouracil Levels as a Diagnostic Marker of Dihydropyrimidine Dehydrogenase Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N16URA
Record Dates: First submitted 2016-02-24; First posted 2016-03-24 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2017-08

CONDITIONS: Drug Safety Biomarkers
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (fasting) (No Intervention): Fasting condition
- B (fed) (Experimental): Fed condition (test meal)
  Interventions: Other: Test meal (breakfast)

INTERVENTIONS:
Other: Test meal (breakfast) — Standardized test meal, in accordance with high-fat and high-calorie meal as described in the FDA guidance, but ingredients are changed to Dutch standards and ingredients are added that are expected to have the largest effects on dihydrouracil and uracil levels
  Arms: B (fed)

SUMMARY:
Healthy volunteer food-effect study to determine the effect of food on uracil and dihydrouracil levels in plasma

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer; not known with cancer or current treatment for cancer
2. Age at least 18 years
3. Able and willing to give written informed consent
4. Able and willing to consume the prescribed breakfast
5. Able and willing to undergo blood sampling

Exclusion Criteria:

1. Any treatment with investigational drugs within 30 days before the start of the study
2. Any condition that may interfere with the study protocol
3. Women who are pregnant
4. Allergies or intolerance for components of the prescribed breakfast

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Uracil levels (ng/ml) and dihydrouracil levels (ng/ml), compared in fed and fasting condition | 2 test days
  12 blood samples taken on both test days (fed and fasting condition), to investigate the effect of food on uracil and dihydrouracil levels

SECONDARY OUTCOMES:
dihydropyrimidine dehydrogenase enzyme activity (nmol/mg*h) | baseline
  Dihydropyrimidine dehydrogenase enzyme activity is assessed at baseline to rule out any potential influence of dihydropyrimidine dehydrogenase deficiency on uracil and dihydrouracil levels

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schellens, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided